CLINICAL TRIAL: NCT00611780
Title: Prospective Randomized Trial On RadiaTion Dose Estimates Of CT AngIOgraphy In PatieNts Scanned With A 100kV Protocol
Acronym: PROTECTION-II
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: PD Dr. Joerg Hausleiter, Deutsches Herzzentrum
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: GE IDE No. R00207
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2008-08-27 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Disease
Keywords: Coronary CT angiography; Radiation dose estimates
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Reduced tube voltage of 100kV.
  Interventions: Radiation: tube voltage
- 2 (Active Comparator): Standard tube voltage of 120kV.
  Interventions: Radiation: tube voltage

INTERVENTIONS:
Radiation: tube voltage — standard 120 kV
  Arms: 2
Radiation: tube voltage — reduced voltage of 100 kV
  Arms: 1

SUMMARY:
The objective of this study is to compare radiation dose of a 100kV scan protocol to the standard 120kV scan protocol. We hypothesize that the 100kV scan protocol is associated with a reduction in dose estimates of at least 20%, while the diagnostic image quality is not inferior.

Secondary endpoints of the study include quantitative image quality parameters, diagnostic accuracy for 120 vs.100kV studies compared to invasive angiography in patients who underwent subsequent invasive coronary angiography

DETAILED DESCRIPTION:
All patients scheduled for a coronary CT scan are screened for inclusion and exclusion criteria. Patients are included if they have stable sinus rhythm (heart rate <100 bpm) and a body weight < 90 kg or a body mass index (BMI) < 30. Informed signed consent is obtained from these patients and the CT scan is prepared. After topogram scan and the native scan for Ca-Scoring, patients are randomized in two groups with the use of sealed envelopes. After that contrast-enhanced coronary CT angiography is performed with the 120kV- or 100kV-protocol.

The CT examination is evaluated by two experienced investigators on a per-vessel basis and all results and study-related data are collected in a dedicated database. For assessment of image quality, a previously established 4-point score system is used and quantitative image quality parameters are measured.

A 30 day follow-up after the CT examination aims to evaluate if patients underwent invasive coronary angiography or were scheduled for a myocardial stress / perfusion test (such as stress-echocardiography, myocardial scintigraphy or stress perfusion imaging by MRI).

ELIGIBILITY:
Inclusion Criteria:

* patients with an indication for a coronary CT angiography (planned evaluation of the coronary arteries)
* stable sinus rhythm
* patient weight < 90kg or body mass index < 30 kg/m2
* signed informed consent

Exclusion Criteria:

* non-ECG triggered studies
* non-coronary CTA studies, e.g. bypass graft CTAs, pre- or post EP studies, CABG planning studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Compared with a 120kV protocol the use of a 100kV scan protocol is associated with a reduction in dose estimates of at least 20%, while the diagnostic image quality is not inferior. | 30 days

SECONDARY OUTCOMES:
impact of the 100kV scan protocol on quantitative image quality parameters, e.g. image noise, signal and contrast intensity, signal- and contrast-to-noise-ratios | 30 days
diagnostic accuracy (sensitivity, specificity as well as positive and negative predictive values) for 120kV vs. 100 kV studies when compared with invasive coronary angiography on a per-vessel based analysis. | 30 days
frequency of non-diagnostic CTA studies when comparing 120kV and 100kV | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Hausleiter, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Germany

REFERENCES:
- [Derived] Hausleiter J, Martinoff S, Hadamitzky M, Martuscelli E, Pschierer I, Feuchtner GM, Catalan-Sanz P, Czermak B, Meyer TS, Hein F, Bischoff B, Kuse M, Schomig A, Achenbach S. Image quality and radiation exposure with a low tube voltage protocol for coronary CT angiography results of the PROTECTION II Trial. JACC Cardiovasc Imaging. 2010 Nov;3(11):1113-23. doi: 10.1016/j.jcmg.2010.08.016. PMID 21070998